CLINICAL TRIAL: NCT03721497
Title: Muscle Strength and -Mass After Bariatric Surgery - a Possible Effect of Testosterone Replacement Therapy? Randomized, Placebo-controlled and Double-blinded Study
Brief Title: Testosterone in Bariatric Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Line Velling Magnussen, Medical Doctor, PhD, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2018-002365-19
Record Dates: First submitted 2018-10-22; First posted 2018-10-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Bariatric Surgery Candidate; Male Hypogonadism; Muscle Loss
MeSH Terms: conditions — Eunuchism; Muscular Atrophy | interventions — testosterone undecanoate

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled and double-blinded study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone Undecanoate (Active Comparator): Inj. Testosterone undecanoat (Nebido®), 1000 mg im preoperative (baseline, weeks 6, 18 and 30 depending on time to surgery) and postoperative (weeks 4, 16, 28, 40)
  Interventions: Drug: Testosterone Undecanoate
- Placebo (Placebo Comparator): Inj. placebo preoperative (baseline, weeks 6, 18 and 30 depending on time to surgery) and postoperative (weeks 4, 16, 28, 40)
  Interventions: Drug: Testosterone Undecanoate

INTERVENTIONS:
Drug: Testosterone Undecanoate — The patients will be randomly assigned to either testosterone or placebo.
  Other Names: Placebo

SUMMARY:
Bariatric surgery is an effective method in the treatment of severe obesity and type 2 diabetes mellitus achieving high remission rates. However, weight loss also causes loss of skeletal muscle and bone mass which at least partly could be prevented by exercise and dietary intervention although the counselling of obese and sedentary individuals in order to increase their physical activity presents a challenge. As up to 78.8% of men undergoing bariatric surgery have low levels of testosterone, testosterone therapy could be considered an attractive alternative or supplement to prevent the immense loss of muscle mass during weight loss. Furthermore, low testosterone levels are associated with sarcopenia, insulin resistance, increased body fat, reduced quality of life, loss of libido and reduced sexual function. The study is a long-term randomized, placebo-controlled trial investigating the effects of testosterone therapy combined with exercise and diet counselling on body composition, components of the metabolic syndrome, hormones, inflammation, sexual function and quality of life before and after weight loss in obese, hypogonadal men undergoing bariatric surgery.

DETAILED DESCRIPTION:
Introduction Obesity, poor physical fitness and low muscular strength are associated with all-cause mortality. Loss of bodyweight is commonly achieved by diet with or without exercise intervention. However, both diet and diet+exercise programs are often followed by weight regain and it is generally difficult to achieve long-term weight loss.

There are many challenges associated with the counselling of obese and sedentary individuals in order to increase their physical activity (PA), and there may be a need for a tight schematic counselling to achieve positive results. Additionally, promoting PA among patients that have undergone bariatric surgery has also shown to be challenging even though PA may be of a great importance regarding several postoperative outcomes. Lifestyle changes following bariatric surgery may be important for the overall effect of the BS in the long term. Therefore, it is vital to find an appropriate and well-suited setting to improve PA among these patients. When structuring PA counselling, the five A´s (Assess, Advise, Agree, Assist, Arrange) might be a helpful tool and it is considered important to engage the patients in PA counselling both before and after the surgery.

Loss of bodyweight reduces morbidity and mortality. Bariatric surgery is the most effective method to treat severe obesity and type 2 diabetes mellitus achieving high remission rates. However, weight loss also decreases skeletal muscle mass which might counterbalance the positive effects of a bariatric surgery since low lean body mass is linked to increased mortality under various circumstances (i.e., heart disease, cancer, burn injuries). Furthermore, a substantial loss of bone mass is seen after bariatric surgery despite weight stability in the second-year post-operative, which could have important clinical implications for long-term skeletal health with increased fracture risk. On the other hand, the loss of muscle and bone mass could merely be a natural adaptation to a lower weight after bariatric surgery. Studies trying to establish whether the loss of muscle mass is disproportionately in patients following bariatric surgery compared to BMI-matched controls are conflicting, showing lower muscle mass in both sexes after surgery compared with their respective matched controls assessed by magnetic resonance imaging in one study whereas another study has shown comparable fat-free mass 24 months post-operative assessed by bioelectric impedance. Currently, there are no effective approaches to prevent the immense loss of muscle and bone mass following bariatric surgery although several approaches can be considered, e.g. exercise and dietary intervention.

Low testosterone levels have been associated with sarcopenia, insulin resistance, increased body fat, reduced quality of life and loss of libido and sexual function. Testosterone therapy increases lean body mass (i.e. muscle mass), improves bone density and decreases fat mass. As up to 78.8% of patients undergoing bariatric surgery suffer from low testosterone levels, testosterone therapy prior to and after bariatric surgery may prevent or reduce the considerable loss of muscle mass during the weight loss period. So far, no studies have evaluated the effect of testosterone therapy combined with exercise and diet counselling on body composition and quality of life in men undergoing bariatric surgery.

Testosterone therapy and cardiovascular risk Studies on cardiovascular risk during testosterone therapy are conflicting. A study in old men with limitations in mobility showed significantly more cardiovascular events during testosterone therapy compared to placebo and the study was ended prematurely. Low HDL levels are linked to an increased morbidity and mortality of cardiovascular disease. A significant small decrease in HDL cholesterol levels in men treated with testosterone was reported in a meta-analysis and a systematic review. However, a large observational study on pooled data in obese, hypogonadal diabetic men during six years of testosterone therapy reported a favorable change in lipid profile along with reduced pulse pressure and reduced arterial stiffness, which are independent risk factors for cardiovascular disease. Another approach in clarifying the effect of testosterone therapy on cardiovascular disease risk is the evaluation of biomarkers for cardiovascular disease during therapy, i.e. soluble Klotho, a protein, which may function as a hormone. Higher levels of soluble Klotho are independently associated with a lower likelihood of having cardiovascular disease. To date, no reports on Klotho have been published in obese patients undergoing bariatric surgery during testosterone therapy.

Few studies have addressed the influence of testosterone therapy on the haemostatic system. Thrombin generation (TG) measures are risk markers of cardiovascular disease and address the composite of multiple factors that influence blood coagulation. One intervention study showed that i.m. testosterone treatment for one year in elderly men with low testosterone levels had no impact on thrombin generation measured at one year. A significant number of patients sustaining venous thrombotic events after initiation of testosterone therapy often had inherited cardiovascular risk factors such as Factor V Leiden, and thrombotic events were primarily observed within the first months of testosterone treatment, suggesting that testosterone therapy triggers cardiovascular events in thrombosis prone individuals. Thus, studies on both the short term and the long term impact of testosterone treatment on the haemostatic system are warranted.

Pseudo-Cushing's syndrome Central obesity results in a cluster of metabolic abnormalities contributing to premature death, so-called Pseudo-Cushing's syndrome. Glucocorticoids regulate adipose-tissue differentiation, function and distribution, and in excess, cause central obesity. To our knowledge, no studies have reported results on levels of cortisol and testosterone before and after bariatric surgery.

3. Trial plan and design General aim To investigate the effect and clinical relevance of testosterone therapy combined with exercise and diet counselling in hypogonadal men undergoing bariatric surgery.

Objectives To evaluate the effect of testosterone therapy combined with exercise and diet counselling on muscle strength, body composition, hormones, components of the metabolic syndrome, inflammation, sexual function, and quality of life after weight loss in obese, hypogonadal men undergoing bariatric surgery.

Perspective The study will investigate whether testosterone therapy can stabilize muscle function, prevent the substantial decrease in muscle mass (lean body mass), and improve components of the metabolic syndrome, inflammation and quality of life in patients after bariatric surgery.

Study design A two centre, randomized, double-blind, placebo-controlled study on testosterone therapy combined with lifestyle intervention, in men eligible for bariatric surgery with low testosterone levels. Routine bariatric procedure will be conducted between 3 and 6 months after inclusion. The end of the study is 52 weeks postoperatively.

Method A randomized, double-blind, placebo-controlled intervention study in men eligible for bariatric surgery and low testosterone levels (total testosterone < 12.0 nmol/l). Routine bariatric procedure will be conducted between 3 and 6 months after inclusion.

4. Study population Recruitment Patients will be recruited among bariatric patients at Hospital of Southwest Jutland and at Odense University Hospital. As part of a review of existing clinical practice in the Region of Southern Denmark, patients who are entitled to bariatric surgery are currently subject to an audit with the establishment of a quality and research database. As part of the audit, patients have had their testosterone levels in the blood measured. The investigators of the study may obtain these results from the journal, if there is a signed consent statement during the audit, where the patients also have agreed to be contacted for future projects. Inclusion will be in the beginning of the mandatory 8% weight loss period lasting 3-6 months.

Randomization After the baseline assessment, the patients will be randomly assigned to either testosterone or placebo. The randomization sequence will be created using OPEN Randomise, stratifying patients with a 1:1 allocation using random block sizes of 2, 4 and 6. The allocation sequence will be concealed from the researcher enrolling and OPEN Randomise will send an e-mail to an email address each time a randomization is performed.

5. Treatment of patients Treatment regimen

* Inj. Testosterone undecanoat (Nebido®), 1000 mg im or placebo preoperative (baseline, weeks 6, 18 and 30 depending on time to surgery) and postoperative (weeks 4, 16, 28, 40) (Table 1).
* Administration: deep and slow (over two minutes) intragluteal injection
* Due to the risk of anaphylaxis, patients are observed at least 30 minutes on the test site after the first two injections

Non-pharmacological intervention

* Routine bariatric procedure (Roux en Y gastric bypass or sleeve gastrectomy). Surgery will be conducted between 3 and 6 months after inclusion.
* Lifestyle intervention program: Routine instructions on diet and dietary precautions after surgery and individual exercise counseling three times after surgery.

Contraindications Testosteron undecanoate (ATC-code G03BA03)

* previously diagnosed with prostate, mammae or liver cancer. Any other cancer within the last 5 years.
* hypersensitivity to the active substance or to any of the excipients Caution in
* cardiac insufficiency, especially known ischemic heart disease and hypertension
* hepatic or renal insufficiency
* clotting disorders / anti-coagulant treatment
* known epilepsy and migraine
* pre-existing sleep apnoea

Study medicine is administered at the departments of endocrinology at SVS. Study medicine is handled according to annex 13.

Patients are treated with Testosterone Undecanoate 1000 mg/4 ml, intramuscular (i.m.) or placebo.

Study medicine and placebo have been produced by Bayer Health Care. Packing, blinding, labeling and randomization of study medicine are done by the pharmacy of Odense University Hospital according to annex 13: Name of sponsor, route of administration, batch number, trial reference code, user manual for study medicine, storage of study medicine expiration date (a copy of the label is placed in the trial master file).

The medicine (active and placebo) is delivered to the pharmacy from Bayer with no labels. Identical labels will be put on the ampules, with the exception of the randomization number.

Study medicine can be used only in clinical trials. Sponsor is responsible for the destruction of surplus medicine.

Discontinuation of study treatment

Treatments stop:

* Confirmed increase in serum PSA > 3 ug/l and clinical symptoms and at least 20% increase since baseline is followed by referral to urological evaluation
* Suspicion of prostate cancer
* Hematocrit (EVF) > 0.52 and at least 20% increase since baseline
* Serum ALAT >3 times upper normal limit and at least 20% increase since baseline
* Patients can leave the study prior to end of study, due to safety issues (increased safety parameters), fulfillment of exclusion criterion, at own request or due to lack of compliance including failure to achieve 8% weight loss prior to operation.

Safety evaluation

Monitoring:

* Physical examination (baseline, per/postoperative weeks 0, 28 and 52) (Table 1)
* Biochemical examinations: 1. testosterone levels (baseline) 2. PSA, EVF, ALAT (baseline, preoperative weeks 6 and 18, postoperative weeks 0, 16, 28 and 52)
* Clinical relevant abnormal measurements are repeated

Safety parameters:

* Measurements of hematocrit: testosterone therapy increases the hematocrit level and high levels of hematocrit leads to higher risks of venous thrombosis (Danish Urological Society (DUS) 2013).
* In order to take into account the Danish Urology Cancer Group (DUCG) 2013 report on prostate cancer, and the Danish Urological Society report on androgen substitution (2013) the exclusion criterion for PSA in the study is based on the above level.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for bariatric surgery according to the Danish national criteria (i.e. aged 18-60 years, BMI >35 kg/m2 with specific secondary disease or BMI >40 kg/m2 with significant health issues assessed by the multidisciplinary bariatric team) [42]
* Caucasian men
* Total testosterone < 12.0 nmol/l
* No contraindications for testosterone treatment

Exclusion Criteria:

* Previously diagnosed with prostate, mammae or liver cancer. Any other cancer within the last 5 years.
* Hypersensitivity to the active substance or to any of the excipients in Nebido®
* Symptomatic heart disease NYHA >2
* Recently thromboembolic disease <3 months
* PSA >4.0 ug/l or PSA>3.0 ug/l and lower urinary tract symptoms
* Disability that severely affect the ability to perform exercise training
* EVF > 52%

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal isometric muscle strength (N) in shoulder muscles | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  shoulder elevation

SECONDARY OUTCOMES:
Change in Lean body mass (kg) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  assessed using Dual x-ray absorptiometry (DEXA) on Hologic Discovery devices (Waltham, MA, US)
Change in Total bone mass and density (BMC and BMD) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Assessed using Dual x-ray absorptiometry (DEXA) on Hologic Discovery devices (Waltham, MA, US)
Change in Total fat mass (kg) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Assessed using Dual x-ray absorptiometry (DEXA) on Hologic Discovery devices (Waltham, MA, US)
Change in BMI (regional body composition) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  weight/height² (kg/m²)
Change in Waist/hip-ratio (regional body composition) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Waist: will be measured in the middle of the distance between the 12th rib and antero-superior iliac spine, while keeping the measuring tape parallel with the floor. Hip: will be measured across the widest part of the hips while keeping the tape parallel to the floor. Hip: will be measured across the widest part of the hips while keeping the tape parallel to the floor. Waist/hip ratio will be computed
Change in Maximal isometric muscle strength in lower extremities (N) (strength) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  hip extension and abduction
Change in Maximal isometric muscle strength in upper extremities (N) (strength) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  shoulder abduction, shoulder adduction
Change in VO2-max | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Maximal oxygen uptake will be estimated from the relation between sub-maximal workload and stable heart rate obtained in Åstrand one-point sub-max test.
Change in stair climb test | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  The outcome is the number of times the subjects are able to reach the stairs up and down for a period of one minute
Change in HOMA-R | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  HOMA1-IR = (fasting plasma insulin (mU/l)xfasting plasma glucose(mmol/l))/22.5
Change in HbA1c (mmol/mol) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Evaluation of glucose metabolism
Change in Fasting-P-Blood glucose (mmol/l) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Evaluation of glucose metabolism
Change in Coagulation/fibrinolysis status | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  thrombin generation measures
Change in Leptin (µg/L) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in Adiponectin (mg/L) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in hsCRP | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in IL-6 | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in suPAR | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in lipid profile: HDL, LDL, triglycerides in mmol/l | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in Cortisol and cortisol metabolites | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  urine sample
Change in Cortisol | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in growth hormone-axis (IGF-I and IGF-II, IGFBPs, bioactive IGF-I) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in soluble Klotho | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in fibulin-1 | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in 1CTP | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in CTX | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in PTH | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in 25OH-vitaminD | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in 1.25(OH)2-Vitamin-D | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in osteocalcin | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in PINP | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  blood sample
Change in International Index of Erectile Function (IIEF-5) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Questionnaire on sexuality
Change in Major Depression Inventory (MDI) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Questionnaire on depression and mental well-being
Change in Short Form 36 (SF-36) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Questionnaire on quality of life
Change in World Health Organization Well Being Index (WHO-5) | At baseline preoperatively and at weeks 0, 28 and 52 per/postoperatively
  Questionnaire on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Line V Magnussen, MD, PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- HospitalSWD, Esbjerg, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT03721497/Prot_SAP_000.pdf